CLINICAL TRIAL: NCT04824586
Title: Intraoperative Insulin Administration (Infusion Regimen vs. Bolus Regimen) at Cardiac Surgery for Type II Diabetic Patients; A Randomised Control Trial.
Brief Title: Intraoperative Insulin Administration at Cardiac Surgery for Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hashemite University (Other)
Responsible Party: Principal Investigator, Mohanad Mousa Taha Odeh, Director of Pharmacy Management & Pharmaceutical Care Innovation Centrer, The Hashemite University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Intraoperative Insulin
Record Dates: First submitted 2021-03-20; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus; Cardiac Event
Keywords: Type II diabetes mellitus; Cardiac surgery; Insulin; Insulin infusion regimen; Insulin bolus regimen
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: This study was a parallel-group, randomized, controlled trial with 1:1 allocation ratio.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin infusion regimen (Experimental): Adult type II diabetic patients, who were admitted to hospital for cardiac surgery. These group received their dose of insulin; Insulin infusion regimen.
  Fast-acting human insulin (Actrapid®) was used in this group.
  Interventions: Drug: Fast-acting human insulin
- Insulin bolus regimen (Experimental): Adult type II diabetic patients, who were admitted to hospital for cardiac surgery. These group received their dose of insulin; Insulin bolus regimen.
  Fast-acting human insulin (Actrapid®) was used in this group.
  Interventions: Drug: Fast-acting human insulin

INTERVENTIONS:
Drug: Fast-acting human insulin — Both patients in the infusion or bolus group received their dose of insulin. The protocol of the insulin regimen and its related details were carried out according to the standard recommendations in a hospital where the trial done.
  Other Names: Actrapid®

SUMMARY:
The primary objective of the study was to explore which insulin-based regimen is better, infusion or bolus regimen, for intraoperative management of glucose level for the diabetic patient at cardiac surgery. Secondary objectives include: comparing the relative amounts of insulin needed during the operation and subsequent cost impact and comparing potassium levels between groups.

Ethical approval for the study was obtained from the Office for Research Ethics Committees at Hashemite University - Prince Hamza hospital.

This study was a parallel-group, randomized, controlled trial with 1:1 allocation ratio.

Participants: Adult diabetic patients, type 2, who were admitted to hospital for cardiac surgery.

The intervention: Both patients in the infusion or bolus group received their dose of insulin, fast-acting human insulin (Actrapid®) was used.

Setting: Patients were recruited at Prince Hamza hospital, Amman, Jordan. A tertiary care center specialized unit in cardiac surgery for diabetic patients.

Outcomes monitoring: It was monitored six times as follows: preoperative induction measure, then glucose post heparin, and after that for 2 hours, glucose levels were monitored every 30 minutes. Insulin quantities were recorded as well to be used in secondary outcomes analysis.

Randomization, allocation, and blinding During patient enrolment, concealed allocation to either infusion group or bolus group was guaranteed through the use of a closed envelope system prepared by an independent investigator. Block randomization with random block sizes, ensured allocation balance, and avoided selection bias by preventing allocation prediction. Researchers and physicians were blind to the block size sequence and randomization. Envelopes were unopened until completion of patient registration. Hospital staff who monitor glucose and those who administered insulin were blinded to the primary and secondary outcomes' measure.

DETAILED DESCRIPTION:
The primary objective of the study was to explore which insulin-based regimen is better, infusion or bolus regimen, for intraoperative management of glucose level for the diabetic patient at cardiac surgery. Secondary objectives include: comparing the relative amounts of insulin needed during the operation and subsequent cost impact and comparing potassium levels between groups.

Ethical approval and study registration Ethical approval for the study was obtained from the Office for Research Ethics Committees at Hashemite University - Prince Hamza hospital with reference number 2/1/2019/2020.

Methods and Materials This study was a parallel-group, randomized, controlled trial with 1:1 allocation ratio.

Participants Adult diabetic patients, type 2, who were admitted to hospital for cardiac surgery. In addition to signing the consent form, patients were recruited when they met the following criteria: >40 years old, patients who need the usual insulin according to insulin dosing guidelines, patients with pre-operation glucose level > 200 mg/dL and < 300 mg/dL.

The following patients were excluded: Insulin sensitive patents (Age >70 years, Glomerular Filtration Rate (GFR) <45 ml/min, No history of Diabetes, Insulin resistance patients (Body Mass Index > 35 kg/m2, total daily insulin dose >80 units, Steroids > 20 mg prednisone daily, patients who at high risk of complications and or (those whom their operation was differed to be supervised by a specialized team). Patients who were unable to give written informed consent, who had ≥4 emergency admissions during the six months prior to the index admission.

The intervention Both patients in the infusion or bolus group received their dose of insulin, fast-acting human insulin (Actrapid®) was used. The protocol of the insulin regimen and its related details were carried out according to the standard recommendations.

Setting Patients were recruited at Prince Hamza Hospital, Amman, Jordan. A tertiary care center specialized unit in cardiac surgery for diabetic patients.

Diabetic patients who had booked cardiac surgery and met the criteria were invited to the study. Patients who accepted participation and signed the consent were recruited by well-trained research assistance, who was trained on an ethical standard and patient-centered approach.

Primary and secondary outcomes In the present study, the primary outcome was the intraoperative level of glucose. It was monitored six times as follows: preoperative induction measure, then glucose post heparin, and after that for 2 hours, glucose levels were monitored every 30 minutes. Insulin quantities were recorded as well to be used in secondary outcomes analysis.

Sample size To detect a difference of at least 25mg/dL between infusion and bolus groups (the standard deviation of the two groups is expected to be 35 mg/dL, i.e., the variance is 1225 mg/dL), the study will need to recruit and record full data for at least 31 patients in each group. Providing that significant level of confidence 95% and the power of 80%.

n = (Zα/2+Zβ)2 *2*σ2 / d2. where Zα/2 is the critical value of the Normal distribution at α/2 (for a confidence level of 95%, α is 0.05, and the critical value is 1.96), Zβ is the critical value of the Normal distribution at β (for a power of 80%, β is 0.2, and the critical value is 0.84), σ2 is the population variance, and d is the difference needed to be detected.

Statistical methods Standard independent-samples t-test or separate variances t-test (Welch t-test) was used to compare the results between the two arms of the study. General Linear Model, one-way repeated measures ANOVA was conducted to determine whether there was a statistically significant difference within groups. Cost analysis and cost-effectiveness were used for the pharmacoeconomic analysis. Incremental cost-effectiveness ratio (ICER) was calculated as the cost of insulin in the Infusion protocol minus the cost of insulin in the bolus protocol divided by drop-in glucose level by infusion - drop in glucose level by bolus).

Randomization, allocation, and blinding During patient enrolment, concealed allocation to either infusion group or bolus group was guaranteed through the use of a closed envelope system prepared by an independent investigator. Block randomization with random block sizes, ensured allocation balance, and avoided selection bias by preventing allocation prediction. Researchers and physicians were blind to the block size sequence and randomization. Envelopes were unopened until completion of patient registration. Hospital staff who monitor glucose and those who administered insulin were blinded to the primary and secondary outcomes' measure.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients, type 2, who were admitted to hospital for cardiac surgery.
* Patient above 40 years old,
* Patients who need the usual insulin according to insulin dosing guidelines
* Patients with pre-operation glucose level > 200 mg/dL and < 300 mg/dL.

Exclusion Criteria:

* Insulin sensitive patents (Age >70 years, Glomerular Filtration Rate (GFR) <45 ml/min, No history of Diabetes, Insulin resistance patients (Body Mass Index > 35 kg/m2, total daily insulin dose >80 units, Steroids > 20 mg prednisone daily, patients who at high risk of complications and or (those whom their operation was differed to be supervised by a specialized team).
* Patients who were unable to give written informed consent.
* Patients have ≥4 emergency admissions during the six months prior to the index admission.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative level of glucose | Change from baseline glucose level (preoperative) at six hours intraoperative
  To explore which insulin-based regimen is better, infusion or bolus regimen, for intraoperative management of glucose level for the diabetic patient at cardiac surgery.

SECONDARY OUTCOMES:
Insulin quantities | Change from baseline glucose level (preoperative) at six hours intraoperative
  To compare the relative amounts of insulin needed during the operation and subsequent cost impact and comparing potassium levels between groups

CONTACTS AND LOCATIONS:
Overall Officials: Mohanad M Odeh, PhD, Principal Investigator — The Hashemite University
Locations (1):
- Prince Hamza Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No